CLINICAL TRIAL: NCT04403659
Title: Monitoraggio Telematico di Pazienti Ricoverati in Ospedalizzazione a Domicilio Per Scompenso Cardiaco Acuto - Studio Pilota
Brief Title: Telemonitoring of Patients Admitted in Hospital at Home With Acute Decompensated Heart Failure - Pilot Study
Acronym: MONTEROSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: Santer Reply S.p.A. Milan, Italy (Unknown); Caretek S.r.l. Turin, Italy (Unknown)
Responsible Party: Principal Investigator, Dott.ssa RENATA MARINELLO, Principal Investigator, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MONTEROSA
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Heart Failure; With Decompensation; Heart Failure，Congestive; Heart Failure Acute
Keywords: Telemedicine; Telemonitoring; Hospital at Home; Home Hospitalization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Use of a telemonitoring/telemedicine suite (including a sphygmomanometer, pulse oximeter, weight scale, thermometer, glucometer, electrocardiograph) as a support to the routine clinical care
  Interventions: Device: Telemedicine/telemonitoring (TM) suite
- Control (No Intervention): Routine clinical care, following European Society of Cardiology 2016 Guidelines on Heart failure and Good Clinical Practice guidelines

INTERVENTIONS:
Device: Telemedicine/telemonitoring (TM) suite — The couples patient/caregiver will receive and trained to use a suite of TM instruments including: sphygmomanometer, pulse oximeter, weight scale, thermometer, glucometer, electrocardiograph. During the intervention phase (i.e. from allocation to exit from the study), the caregiver/patient will be asked to measure twice daily, at prespecified times, the following parameters using TM devices: arterial blood pressure, peripheral arterial haemoglobin saturation, tympanic temperature. Body weight will be evaluated once daily.
  The TM glucometer and TM electrocardiograph will be used exclusively by healthcare staff in case of patients in need of capillary blood glucose testing and according to clinical needs, respectively. All data will be automatically sent to a central interface and made readily available to physicians and nurses, to enable a prompt clinical response. In case of malfunctioning, a technical support will be ensured.
  Arms: Intervention

SUMMARY:
"La Casa nel Parco" (CANP) Project is a multidisciplinary project funded by the European Union and Regione Piemonte aimed to explore innovative technology application in the care of older subjects. In this context, MONTEROSA is a monocentric randomized controlled open-label clinical trial evaluating the use of a telemonitoring/telemedicine (TM) suite (including a sphygmomanometer, pulse oximeter, weight scale, thermometer, glucometer, electrocardiograph) as a support to the routine clinical care of patients admitted to a Hospital at Home service for acute decompensated heart failure.

The main objective of the study will be to evaluate the impact of TM on number of daily physician's visits. Secondary objectives will be to evaluate the impact of TM on number of daily nurse visits, on overall in-hospital mortality and on patient's and caregiver's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in Hospital at Home with signs and/or symptoms of new-onset or decompensated heart failure, according with the definition of 2016 European Society of Cardiology (ESC) guidelines on Heart Failure
* Written informed consent signed by both the patient and the main caregiver

Exclusion Criteria:

* Main caregiver with low IT skills (e.g. unable to use a smartphone);
* Patient in whom body weight or accurate daily urine output cannot be measured
* Patient with history of neoplastic/degenerative disease and with estimated life expectancy less than 3 months
* Patient with decompensated liver cirrhosis (Child-Pugh score B o C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Mean daily number of physician visits | From allocation through to HaH discharge, in mean 15 days
  Mean daily number of physician visits during Hospital at Home (HaH) stay, defined as total number of physician visits during HaH stay, divided by days of HaH stay, for every single patient

SECONDARY OUTCOMES:
Mean daily number of nurse visits | From allocation through to HaH discharge, in mean 15 days
  Mean daily number of nurse visits during Hospital at Home (HaH) stay, defined as total number of nurse visits during HaH stay, divided by days of HaH stay, for every single patient
Mean daily number of urgent physician visits | From allocation through to HaH discharge, in mean 15 days
  Mean daily number of urgent physician visits during Hospital at Home (HaH) stay, defined as total number of urgent (i.e. unplanned) physician visits during HaH stay, divided by days of HaH stay, for every single patient
Mean daily number of urgent nurse visits | From allocation through to HaH discharge, in mean 15 days
  Mean daily number of urgent nurse visits during Hospital at Home (HaH) stay, defined as total number of urgent (i.e. unplanned) nurse visits during HaH stay, divided by days of HaH stay, for every single patient
Overall mortality | From allocation through to HaH discharge, in mean 15 days
  Death by any cause during Hospital at Home (HaH) stay
Patient's quality of life evaluated through the 12-Item Short Form survey (SF-12) | At HaH discharge, in mean 15 days after allocation
  Patient's quality of life evaluated through the 12-Item Short Form survey (SF-12), stratified in Physical component summary (Pcs) and Mental component summary (Mcs), at Hospital at Home (HaH) discharge
Main caregiver's quality of life evaluated through the 12-Item Short Form survey (SF-12) | At patient's HaH discharge, in mean 15 days after allocation
  Main caregiver's quality of life evaluated through the 12-Item Short Form survey (SF-12), stratified in Physical component summary (Pcs) and Mental component summary (Mcs), at Hospital at Home (HaH) discharge

CONTACTS AND LOCATIONS:
Overall Officials: Renata Marinello, MD, PhD, Principal Investigator — OAU Città della Salute e della Scienza di Torino, Turin, Italy
Locations (1):
- S.C. Geriatria e Malattie Metaboliche dell'Osso U, A.O.U. Città della Salute e della Scienza di Torino, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tibaldi V, Isaia G, Scarafiotti C, Gariglio F, Zanocchi M, Bo M, Bergerone S, Ricauda NA. Hospital at home for elderly patients with acute decompensation of chronic heart failure: a prospective randomized controlled trial. Arch Intern Med. 2009 Sep 28;169(17):1569-75. doi: 10.1001/archinternmed.2009.267. PMID 19786675
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042